CLINICAL TRIAL: NCT01321697
Title: A Non-Randomized Study to Evaluate Leg Lymphatic Drainage Associated With Surgical Intervention for Vulvar Cancer
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator Request
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Other Study IDs: 110583
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Vulvar Cancer
Keywords: Being seen in the Winthrop P. Rockefeller Cancer Institute for vulvar; cancer requiring lymph node evaluation for the ipsilateral or contralateral; groin
MeSH Terms: conditions — Vulvar Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vulvar Cancer
  Interventions: Procedure: Routine Leg edema and groin dissection

INTERVENTIONS:
Procedure: Routine Leg edema and groin dissection — The investigators will be documenting and reporting the variations in leg lymphatic drainage sentinel lymph node biopsy with inguinal-femoral lymph node dissection.

SUMMARY:
This will be a non-blinded, non-randomized study to further our knowledge of and experience with lymph node surgery. The investigators are interested in documenting and reporting the variations in leg lymphatic drainage sentinel lymph node biopsy (SLNB) with inguinal-femoral lymph node dissection (IFLND). The study will be open at the Winthrop P. Rockefeller Cancer Institute at The University of Arkansas for Medical Sciences (UAMS). Dr. Pamela Stone, Dr.Alexander Burnett, and Dr. Juan Roman will be responsible for accruing subjects to this study. It will be open to all patients presenting to the Winthrop P. Rockefeller Cancer Institute with vulvar cancer requiring lymph node evaluation for the ipsilateral and/or contralateral groin who have not had prior groin surgery or radiation to the groins. Patients must meet inclusion and exclusion criteria to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18-100 years of age.
* All races and ethnicities.
* Being seen in the Winthrop P. Rockefeller Cancer Institute for vulvar cancer requiring lymph node evaluation for the ipsilateral or contralateral groin.
* Willing participation following informed consent process.

Exclusion Criteria:

* Has not had prior groin surgery or radiation to the groins.
* Any condition the PI or study physician determines that will put the subject at risk during the procedure.
* Allergy to blue dye used in lymphatic identification.
* Pregnant or breast feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Gynecology Oncology Clinic
Sampling Method: Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vulvar Cancer: Routine Leg edema and groin dissection : The investigators will be documenting and reporting the variations in leg lymphatic drainage sentinel lymph node biopsy with inguinal-femoral lymph node dissection.
Period: Overall Study
Arm/Group | Vulvar Cancer
Started | 7
Completed | 0
Not Completed | 7
Not completed — Study Terminated | 7

BASELINE CHARACTERISTICS:
Arm/Group | Vulvar Cancer
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Successful Identification of Vulvar Sentinel Lymph Nodes Via Gamma Probe.
Time Frame: at time of surgery
Population: Data were not collected/analyzed due to study termination.
Arm/Group | Vulvar Cancer
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Vulvar Cancer
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
Early termination of the study due to investigator decision. No subjects were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes